CLINICAL TRIAL: NCT06438809
Title: Safety and Preliminary Efficacy of Umbilical-Cord-Derived Mesenchymal Stem Cells Injection for Chronic Radiation Proctitis
Brief Title: Umbilical-Cord-Derived Mesenchymal Stem Cells Injection for Chronic Radiation Proctitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-SC01-RP-I/II-03
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic Radiation Proctitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label single arm study (Experimental): All patients will receive a single injection of umbilical cord-derived mesenchymal stem cells (120 million cells), and their therapeutic response will be monitored over a period of 24 months.
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — MSC suspension single does injection.

SUMMARY:
A Phase I/II study to evaluate the safety and preliminary efficacy of human umbilical cord-derived mesenchymal stem cell injection for the treatment of chronic radiation proctitis.

DETAILED DESCRIPTION:
Radiation therapy is frequently used to treat pelvic cancers such as anal, cervical, prostate, and rectal cancer. While effective in controlling local tumors, it can also cause collateral damage to the gastrointestinal tract. The rectum is particularly vulnerable to radiation damage due to its fixed position in the pelvis. In the acute phase, radiation can lead to proctitis, an inflammatory condition characterized by mucosal ulceration, edema, and loss of microvilli. Patients typically present within three months of radiation therapy with symptoms like diarrhea, urgency, and tenesmus. Chronic radiation proctitis can either follow the acute phase or appear after a symptom-free period, typically 8 to 12 months post-radiation treatment. This chronic condition results from radiation-induced small-vessel injury, causing ischemia, obliterative endarteritis, fibrosis, and neovascularization. Rectal bleeding is a common symptom of chronic radiation proctitis.

Clinical studies have demonstrated that mesenchymal stem cell (MSC) treatment offers significant benefits, including anti-inflammatory, immune modulation, and tissue repair effects. Recent research indicates that intralesional injection of MSC is effective in treating radiation proctitis, reducing pain and bleeding without causing severe adverse events. This suggests that MSC treatment could be a promising option for radiation proctitis.

This is a phase I/II study designed to evaluate the safety and preliminary efficacy of MSC treatment for radiation proctitis. Patients will be followed up for 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and sign the informed consent form;
2. Age ≥18 years and <80 years;
3. Good physical condition (WHO performance status score 0-1);
4. Pathologically diagnosed with pelvic malignant tumors and received radiotherapy;
5. Diagnosed with chronic radiation proctitis after at least 6 months of endoscopic examination following the completion of radiotherapy and ineffective conventional treatment;
6. Screening period LENT-SOMA score ≥1;
7. Subjects and their spouses or partners have no plans for conception from screening to 6 months after the end of the trial, no plans for sperm or egg donation, and agree to use effective non-pharmacological contraceptive measures during the trial.

Exclusion Criteria:

1. Patients with severe liver or kidney dysfunction during the screening period;
2. Patients with severe congestive heart failure or coronary artery disease during the screening period;
3. Patients with allergic constitution or severe systemic immune diseases;
4. Patients with active gastrointestinal bleeding or acute intestinal obstruction during the screening period;
5. Pregnant patients;
6. Patients with rectal stenosis or fistula formation requiring surgical treatment that limits endoscopic therapy;
7. Patients with a screening period LENT-SOMA score of 4;
8. Patients with tumor recurrence or metastasis;
9. Patients currently participating in other clinical trials at the time of screening or who have not been out of another clinical trial for less than 1 month;
10. Other situations deemed unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The severity of adverse events after administration as assessed by CTCAE v5.0. | 28 days (1 month)
  Adverse events are any unexpected medical occurrences in a participant that may not be directly caused by the trial intervention. Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 is a grading scale which can be utilized for adverse event (AE) reporting. It ranges from grade 1 (mild) to grade 5 (death related to AE) , and higher grade means the AE is more severe.
The incidence of adverse events after administration. | 28 days (1 month)
  Adverse events are any unexpected medical occurrences in a participant that may not be directly caused by the trial intervention.

SECONDARY OUTCOMES:
The severity of adverse events after administration as assessed by CTCAE v5.0. | 112 days (4 month)
  Adverse events are any unexpected medical occurrences in a participant that may not be directly caused by the trial intervention. Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 is a grading scale which can be utilized for adverse event (AE) reporting. It ranges from grade 1 (mild) to grade 5 (death related to AE) , and higher grade means the AE is more severe.
The incidence of adverse events after administration. | 112 days (4 month)
  Adverse events are any unexpected medical occurrences in a participant that may not be directly caused by the trial intervention.
The recurrence of chronic radiation proctitis symptoms after administration. | Day 112 (month 4)
  The recurrence means that subjects who were previously cured or relieved are diagnosed again by the investigator, clinically, as having chronic radiation proctitis.
The deterioration of chronic radiation proctitis symptoms after administration. | Day 112 (month 4)
  The deterioration means that the symptoms of chronic radiation proctitis have worsened compared to baseline.
No improvement of chronic radiation proctitis symptoms after administration as assessed by LENT-SOMA score. | Day 112 (month 4)
  The Late Effects Normal Tissue/Subjective Objective Management Analytic (LENT/SOMA) is used for grading radiation therapy (RT)-induced side effects. It is graded on a 4-point scale ranging from occasional (score of 1) to refractory (score of 4), with a higher score indicating more severe disease. No improvement means no improvement of the score comparing to the baseline level.
No improvement of chronic radiation proctitis symptoms after administration as assessed by VRS. | Day 112 (month 4)
  The Vienna Rectoscopy Score (VRS) is a feasible and effective tool for detecting and classifying pathological changes in the rectal mucosa after radiotherapy (RT). It is graded on a 5-point scale, ranging from 0 to 5, with a higher score indicating more severe disease. No improvement means that the score does not improve compared to the baseline level.
No improvement of chronic radiation proctitis symptoms after administration as assessed by a semi-quantitative scoring system for radiotherapy-induced rectal pathological damage. | Day 112 (month 4)
  A specific scoring system that assesses the intensity of morphological features has been developed. The total score ranging from 0 to 10 , and a higher score indicates more severe disease. No improvement means that the score does not improve compared to the baseline level.
No improvement of chronic radiation proctitis symptoms after administration as assessed by a RTD grading scale. | Day 112 (month 4)
  The rectal telangiectasia density (RTD) grading scale ranges from 0 to 3, and a higher score indicates the disease is more severe. No improvement means that the score does not improve compared to the baseline level.
No improvement of chronic radiation proctitis symptoms after administration as assessed by VAS score. | Day 112 (month 4)
  The Visual Analogue Scale (VAS) is commonly used to assess the intensity of a patient's pain, ranging from none to extreme. It is graded on an 11-point scale,ranging from 0 to 10,with higher scores indicating more severe pain. No improvement means that the score does not improve compared to the baseline level.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No